CLINICAL TRIAL: NCT02584855
Title: A Phase 3, Multicenter Study With a 36-Week Open-Label Period Followed by a Randomized Double-Blind Withdrawal Period From Week 36 to Week 104 to Evaluate the Long-Term Efficacy and Safety of Ixekizumab (LY2439821) 80 mg Every 2 Weeks in Biologic Disease-Modifying Antirheumatic Drug-Naive Patients With Active Psoriatic Arthritis
Brief Title: A Long-Term Efficacy and Safety Study of Ixekizumab (LY2439821) in Participants With Active Psoriatic Arthritis
Acronym: SPIRIT P3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14518; I1F-MC-RHBF (Other: Eli Lilly and Company); 2015-002433-22 (EudraCT Number)
Record Dates: First submitted 2015-10-16; First posted 2015-10-23 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2018-11

CONDITIONS: Psoriatic Arthritis
Keywords: Spondyloarthritis; Spondylarthropathy
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylarthritis; Spondylarthropathies | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ixekizumab Open Label (Experimental): Open-Label Treatment Period: Starting dose of 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline (week 0) followed by 80 mg given as one SC injection every two weeks (Q2W) from week 2 to randomization (week 36 to 64).
  Interventions: Drug: Ixekizumab
- Ixekizumab (Experimental): Participants completed open label and met criteria for randomization to the double-blind Withdrawal Period.
  Double-Blind Withdrawal Period: 80 mg ixekizumab given as one SC injection Q2W from randomization to week 104 (or, early termination or relapse).
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Participants completed open label and met criteria for randomization to the double-blind Withdrawal Period.
  Double-Blind Withdrawal Period: Placebo given as one SC injection Q2W any time from randomization to week 104 (or, early termination or relapse)
  Interventions: Drug: Ixekizumab; Drug: Placebo
- IXE80Q2W Non-randomized (Experimental): Participants completed open label but did not meet criteria for randomization to the double-blind Withdrawal Period.
  Participants continued to receive 80 mg given as one SC injection every two weeks during the double-blind withdrawal period.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and long-term efficacy of ixekizumab compared to placebo in participants with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Presents with established diagnosis of active psoriatic arthritis (PsA) for at least 6 months, and currently meets Classification for Psoriatic Arthritis (CASPAR) criteria
* Active PsA defined as the presence of at least 3 tender and at least 3 swollen joints
* Presence of active psoriatic skin lesion or a history of plaque psoriasis (Ps)
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment
* Have been treated with 1 or more conventional disease-modifying antirheumatic drugs (cDMARDs)

Exclusion Criteria:

* Current or prior use of biologic agents for treatment of Ps or PsA
* Inadequate response to greater than or equal to 4 conventional disease-modifying antirheumatic drugs (DMARDS)
* Current use of more than one cDMARDs
* Diagnosis of active inflammatory arthritic syndromes or spondyloarthropathies other than PsA
* Have received treatment with interleukin (IL) -17 or IL12/23 targeted monoclonal antibody (MAb) therapy
* Serious disorder or illness other than psoriatic arthritis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (87):
- United States (22):
  - Arizona Arthritis & Rheumatology Research, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis Research, PLC, Phoenix, Arizona
  - University of California, Davis - Health Systems, Sacramento, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Arthritis & Osteoporosis Treatment Center, PA, Orange Park, Florida
  - Florida Medical Clinic PA, Zephyrhills, Florida
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Glacier View Research Institute, Kalispell, Montana
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Weill Cornell Physicians at Brooklyn Heights, Brooklyn, New York
  - Robert A. Harrell, III, MD, Durham, North Carolina
  - Pennsylvania Regional Center for Arthritis & Osteoarthritis, Wyomissing, Pennsylvania
  - Pioneer Research Solutions, Cypress, Texas
  - Arthritis Care & Diagnostic Center P.A., Dallas, Texas
  - Kadlec Clinic Rheumatology, Kennewick, Washington
  - Seattle Rheumatology Associates, P.L.L.C., Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
- Bulgaria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rousse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
- Czechia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Česká Lípa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Praha 4 Nusle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zlín
- Estonia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tartu
- Mexico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuautitlán Izcalli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Poland (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nowa Sól
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nowy Duninów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sochaczew
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yekaterinburg
- Slovakia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Považská Bystrica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Senica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stará Ľubovňa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Svidník
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trnava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zvolen
- South Africa (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempton Park
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Elizabeth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Ukraine (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaporizhzhia
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goodmayes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harlow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Truro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Deodhar AA, Combe B, Accioly AP, Bolce R, Zhu D, Gellett AM, Sprabery AT, Burmester GR. Safety of ixekizumab in patients with psoriatic arthritis: data from four clinical trials with over 2000 patient-years of exposure. Ann Rheum Dis. 2022 Jul;81(7):944-950. doi: 10.1136/annrheumdis-2021-222027. Epub 2022 Apr 7. PMID 35393269
- [Derived] Coates LC, Pillai SG, Tahir H, Valter I, Chandran V, Kameda H, Okada M, Kerr L, Alves D, Park SY, Adams DH, Gallo G, Hufford MM, Hojnik M, Mease PJ, Kavanaugh A; SPIRIT-P3 Study Group. Withdrawing Ixekizumab in Patients With Psoriatic Arthritis Who Achieved Minimal Disease Activity: Results From a Randomized, Double-Blind Withdrawal Study. Arthritis Rheumatol. 2021 Sep;73(9):1663-1672. doi: 10.1002/art.41716. Epub 2021 Aug 6. PMID 33682378
- [Derived] Combe B, Rahman P, Kameda H, Canete JD, Gallo G, Agada N, Xu W, Genovese MC. Safety results of ixekizumab with 1822.2 patient-years of exposure: an integrated analysis of 3 clinical trials in adult patients with psoriatic arthritis. Arthritis Res Ther. 2020 Jan 21;22(1):14. doi: 10.1186/s13075-020-2099-0. PMID 31964419
- See also: Click here for more information about this study: A Long-Term Efficacy and Safety Study of Ixekizumab (LY2439821) in Participants With Active Psoriatic Arthritis (SPIRIT P3) — http://www.lillytrialguide.com/EN/studies/arthritis/rhbf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had four periods: Period 1: Screening period lasting from 4 to 30 days before Week 0, Period 2: Initial open-label treatment period from Week 0 up to Week 36, Period 3: randomized double-blind withdrawal period from Week 36 to week 104 (or, early termination or relapse) and Period 4: post treatment follow-up.
Pre-assignment Details: Participants were randomized during week 36 to week 64. The criteria for randomization in period 3 was having received ixekizumab (IXE) 80 mg Q2W for at least 6 months and meeting Coates criteria for minimal disease activity (MDA) for 3 consecutive months over 4 consecutive visits.The criteria was met anytime from 36 to 64 weeks.
Groups:
- Ixekizumab Open Label: Open-Label Treatment Period (OLTP): Starting dose of 160 milligrams (mg) ixekizumab given as two subcutaneous (SC) injections at baseline (Week 0) followed by 80 mg given as one SC injection every two weeks (Q2W) from week 2 to randomization (week 36 to 64).
- IXE80Q2W Post-Treatment Follow-up Period: Participants did not receive any study treatment during post treatment follow-up period. Post-Treatment Follow-up Period was summarized by last treatment assigned to a participant prior to entering the post-treatment follow up period.
- Placebo Post-Treatment Follow-up Period: Participants did not receive any study treatment during post treatment follow-up period. Placebo Post-Treatment Follow-up Period was summarized by last treatment assigned to a participant prior to entering the post-treatment follow up period.
Period: Open-Label Treatment Period
Arm/Group | Ixekizumab Open Label | IXE80Q2W Non-randomized | Ixekizumab | Placebo | IXE80Q2W Post-Treatment Follow-up Period | Placebo Post-Treatment Follow-up Period
Started | 394 | 0 (Participants completed Open-Label Treatment Period.) | 0 (Participants were randomized to this arm during double-blind withdrawal period.) | 0 (Participants were randomized to this arm during double-blind withdrawal period.) | 0 | 0
Received at Least One Dose of Study Drug | 394 | 0 | 0 | 0 | 0 | 0
Met Randomization Criteria | 158 | 0 | 0 | 0 | 0 | 0
Non-randomized | 133 | 0 | 0 | 0 | 0 | 0
Completed | 291 | 0 | 0 | 0 | 0 | 0
Not Completed | 103 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 61 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — No PI Available | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Withdrawal Period
Arm/Group | Ixekizumab Open Label | IXE80Q2W Non-randomized | Ixekizumab | Placebo | IXE80Q2W Post-Treatment Follow-up Period | Placebo Post-Treatment Follow-up Period
Started | 0 | 133 (Participants completed open label but did not meet criteria for double-blind withdrawal period.) | 79 (Participants completed open label and met criteria for double-blind withdrawal period.) | 79 (Participants completed open label and met criteria for double-blind withdrawal period.) | 0 | 0
Relapsed | 0 | 0 | 67 | 30 | 0 | 0
Completed | 0 | 118 | 77 | 78 | 0 | 0
Not Completed | 0 | 15 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 10 | 0 | 0 | 0 | 0
Not completed — Declined Transfer to a Different Site | 0 | 1 | 0 | 0 | 0 | 0
Period: Post Treatment Follow-up Period
Arm/Group | Ixekizumab Open Label | IXE80Q2W Non-randomized | Ixekizumab | Placebo | IXE80Q2W Post-Treatment Follow-up Period | Placebo Post-Treatment Follow-up Period
Started | 0 | 0 | 0 | 0 | 355 | 12
Completed | 0 | 0 | 0 | 0 | 347 | 12
Not Completed | 0 | 0 | 0 | 0 | 8 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 7 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | Ixekizumab Open Label
Number analyzed (Participants) | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212
  Male | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 330
  Unknown or Not Reported | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 385
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
  Czechia | 90
  Ukraine | 43
  Poland | 60
  Mexico | 16
  South Africa | 26
  United Kingdom | 23
  Slovakia | 16
  Bulgaria | 20
  Estonia | 47
  Russia | 10
  Spain | 11

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Withdrawal Period: Time to Relapse (No Longer Meeting Coates Criteria for Minimal Disease Activity [MDA])
Description: Relapse is loss of MDA response. MDA is achieved if 5 of 7 outcome measures are fulfilled:TJC ≤1;SJC ≤1;psoriasis activity & severity index(PASI total score) ≤1 or body surface area(BSA) ≤3;participant pain VAS score of ≤15;participant global disease activity VAS score of ≤20;HAQ-DI score ≤0.5;and tender entheseal points ≤1.Participants met the randomization criteria if they had MDA for 3 consecutive months over 4 consecutive visits.Time-to relapse was calculated in weeks as follows:((Date of Relapse) - Date of first injection of randomized study treatment in period 3)+1) divided by 7.If the date of first dose is missing,the date of randomization will be used.Participants completing Period 3 will be censored at date of completion(the date of the last scheduled visit in the period).Participants without a date of completion or discontinuation for Period 3 will be censored at latest non-missing date out of the following dates:date of last dose & date of last attended visit in Period 3.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in randomized withdrawal Intent-to-Treat population. Censored participants were Ixekizumab = 49 and Placebo =12.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 79 | 79
Weeks | NA [64.29 to NA] — Median and upper confidence interval could not be estimated due to insufficient events in analysis duration. | 22.29 [16.14 to 28.29]
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Log Rank Test adjusting for geographic region and conventional disease-modifying antirheumatic drug (cDMARD) use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

2. Secondary Outcome: Double-Blind Withdrawal Period: Percentage of Participants Who Relapse in MDA
Description: Relapsed participants are defined as participants no longer meeting Coates criteria for MDA. MDA is achieved if 5 of 7 outcome measures are fulfilled: TJC ≤1; SJC ≤1; psoriasis activity and severity index (PASI total score) ≤1 or body surface area (BSA) ≤3; participant pain VAS score of ≤15; participant global disease activity VAS score of ≤20; HAQ-DI score ≤0.5; and tender entheseal points ≤1.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in randomized withdrawal Intent-to-Treat population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 79 | 79
percentage of participants | 40.5 [29.7 to 51.3] | 86.1 [78.4 to 93.7]
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Logistic regression adjusting for treatment, geographic region, and cDMARD use at the time of double-blind randomization; Test type: Superiority; Odds Ratio (OR) = -45.6, 95% CI 2-sided [-58.8 to -32.3]

3. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Tender Joint Count 68 (TJC)
Description: TJC is the number of tender and painful joints determined for each participant by examination of 68 joints.TJC possible values range from 0 to 68. A lower TJC indicated less number of joints with tenderness. A higher TJC indicated more joint tenderness. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy.
  Loss of Response = Not Meeting less than or equal to 1 TJC. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat Population who had tender joint counts <= 1 at time of randomization. Censored participants: Ixekizumab= 29 and Placebo= 16.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 56 | 57
weeks | 64.29 [24.14 to NA] — Upper confidence interval could not be estimated due to insufficient events in analysis duration. | 22.29 [12.29 to 28.71]

4. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Swollen Joint Count 66 (SJC)
Description: SJC is the number of swollen joints determined for each participant by examination of 66 joints. SJC possible values range from 0 to 66. A lower SJC indicated less joints with swelling. A higher SJC indicated more joints with swelling. Swelling was defined as palpable fluctuating synovitis of the joint.
  Loss of Response = Not Meeting less than or equal to 1 SJC. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat population who had swollen joint counts <= 1 at time of randomization. Censored participants: Ixekizumab= 61 and Placebo = 40.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 72 | 73
weeks | NA [NA to NA] — Median and Confidence interval could not be estimated due to insufficient events in analysis duration. | 28.71 [20.14 to NA] — Upper confidence interval could not be estimated due to insufficient events in analysis duration.

5. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Psoriasis Area and Severity Index (PASI)
Description: The PASI is an index that combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease.
  Loss of Response = Not Meeting less than or equal to 1 PASI total score. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal intent-to-treat population Who had PASI <= 1 at time of randomization. Censored participants: Ixekizumab = 64 and Placebo = 43.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 73 | 77
weeks | NA [NA to NA] — Median and Confidence Interval could not be estimated due to insufficient events in analysis duration. | 36.00 [24.14 to 48.14]
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Log Rank Test adjusting for geographic region and cDMARD use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

6. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: BSA
Description: BSA is an investigator evaluated measure, where the percentage of involvement of psoriasis on each participant's BSA is assessed. BSA was measured on a continuous scale from 0% = no involvement to 100% = full involvement, where 1% corresponded to the size of the participant's handprint including the palm, fingers, and thumb. Loss of Response = Not meeting less than or equal to 3% BSA.
  Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized Withdrawal Intent-to-Treat Population who had BSA <= 3% at time of randomization. Censored participants: Ixekizumab=70 and Placebo= 59.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 73 | 78
weeks | NA [NA to NA] — Median and Confidence Interval could not be estimated due to insufficient events in analysis duration. | NA [36.00 to NA] — Confidence Interval could not be estimated due to insufficient events in analysis duration.
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Log Rank Test adjusting for geographic region and cDMARD use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

7. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Pain Visual Analog Scale (VAS) Score
Description: The pain VAS is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. The VAS contains a continuous line between two endpoints whereby the respondent places a mark on the line to indicate his or her response The scale ranges from 0 (no pain) to 100 (unbearable pain). The scores were measured to the nearest millimeter from the left. Loss of Response = Not Meeting less than or equal to 15 Pain VAS. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat Population who had Pain VAS <= 15 at time of randomization. Censored participants: Ixekizumab=42 and Placebo= 7.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 72 | 68
weeks | NA [36.14 to NA] — Confidence Interval could not be estimated due to insufficient events in analysis duration. | 16.14 [12.14 to 22.71]
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Log Rank Test adjusting for geographic region and cDMARD use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

8. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Patients Global Assessment of Disease Activity (PatGA) Visual Analog Scale (VAS) Score
Description: Participants scored their overall assessment of their psoriatic arthritis (PsA) activity on a 0 to 100 mm horizontal VAS. The scale ranged from 0 (no disease activity) to 100 (extremely active disease activity). The scores were measured to the nearest millimeter from the left.
  Loss of Response = Not Meeting less than or equal to 20 PatGA. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat population Who had PatGA VAS <= 20 at time of randomization. Censored participants: Ixekizumab= 57 and Placebo=18.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 77 | 74
weeks | NA [NA to NA] — Median and Confidence Interval could not be estimated due to insufficient events in analysis duration. | 20.57 [16.14 to 28.14]
Statistical Analysis 1: Comparison: Ixekizumab; Log Rank Test adjusting for geographic region and cDMARD use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

9. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (severe disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
  Loss of Response = Not Meeting less than or equal to 0.5 HAQ-DI. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat population Who had HAQ-DI <= 0.5 at Time of randomization. Censored participants: Ixekizumab= 55 and Placebo=53.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 69 | 68
weeks | NA [NA to NA] — Median and Confidence Interval could not be estimated due to insufficient events in analysis duration. | NA [48.14 to NA] — Median and Upper Confidence Interval could not be estimated due to insufficient events in analysis duration.
Statistical Analysis 1: Comparison: Ixekizumab vs Placebo; Log Rank Test adjusting for geographic region and cDMARD use at the time of double blind randomization; Test type: Superiority; p < 0.001, Log Rank

10. Secondary Outcome: Double-Blind Withdrawal Period: Time to Loss of Response in Each Individual Component of MDA: Tender Entheseal Points
Description: Tender entheseal points was based on the assessment of the 18 entheseal points. Loss of Response = Not Meeting less than or equal to 1 Tender Entheseal Point. Time to loss of response (in weeks) = (date of loss of response - date of first injection of randomized dose of study treatment in the Randomized Double-Blind Withdrawal Period + 1)/7.
Time Frame: Double Blind Randomization through Week 104 (or Early Termination or Relapse)
Population: All participants who received at least one dose of study drug in the randomized withdrawal Intent-to-Treat Population who had tender Entheseal Point <= 1 at time of randomization. Censored participants: Ixekizumab= 58 and Placebo= 58.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Placebo: Double-Blind Withdrawal Period: Placebo given as one SC injection Q2W any time from randomization to week 104 (or, early termination or relapse).
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 73 | 72
weeks | NA [NA to NA] — Median and Confidence Interval could not be estimated due to insufficient events in analysis duration. | NA [60.29 to NA] — Median and Upper Confidence Interval could not be estimated due to insufficient events in analysis duration.

11. Secondary Outcome: Open-Label Treatment Period: Time to Achieve Randomization Criteria (Meeting MDA for 3 Consecutive Months Over 4 Consecutive Visits)
Description: Time to meeting MDA for 3 Consecutive Months Over 4 Consecutive Visits. Time to first response (in weeks) = [(date of first response - date of first injection of study treatment in the Open-Label Treatment Period)+1]/7.
  Open-Label Treatment Period ended at the time when a participant was randomized so the end time was not the same for all participants. Participants were randomized only if they met randomization criteria which was at anytime from week 36 to week 64.
Time Frame: Open Label Baseline through Double-Blind Randomization (Week 36 to 64)
Population: All participants who received at least one dose of study drug in initial open-label treatment period. Censored participants were 239.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab Open Label
Number analyzed (Participants) | 394
weeks | 64.43 [56.14 to NA] — Upper confidence interval could not be estimated due to insufficient events in analysis duration.

12. Secondary Outcome: Double-Blind Withdrawal Period: Time to Re-Gain MDA Following Relapse in MDA
Description: MDA is achieved if 5 of 7 outcome measures are fulfilled: TJC ≤1; SJC ≤1; psoriasis activity and severity index (PASI total score) ≤1 or BSA ≤3; participant pain VAS score of ≤15; participant global disease activity VAS score of ≤20; HAQ-DI score ≤0.5; and tender entheseal points ≤1. Time to first response (in weeks) = (date of first response - date of first injection of study treatment in the Relapse Period + 1)/7.
Time Frame: Relapse in MDA After Double Blind Randomization through Week 104 (or Early Termination)
Population: All participants who received at least one dose of study drug and relapsed in MDA After Double Blind Randomization Until Re-Gain MDA. Censored participants were: Ixekizumab= 3 and Placebo= 3.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 30 | 67
weeks | 4.71 [4.14 to 8.29] | 4.14 [4.14 to 4.29]

13. Secondary Outcome: Double-Blind Withdrawal Period: Change From Baseline in Physical Functioning Assessed by the Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (severe disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.Least Square (LS) mean calculated using Mixed Model Repeated Measurements (MMRM) analysis with treatment group, baseline measure, geographic region, cDMARD use, treatment week, baseline measure-by-treatment week interaction term, and treatment week-by-treatment interaction term as fixed factors.
  Participants were randomized only if they met randomization criteria which was at anytime from week 36 to week 64.
Time Frame: Baseline, 40 Weeks from Double Blind Randomization (Week 36 to 64)
Population: All participants who received at least one dose of study drug had a baseline and post baseline measure in the Double-Blind Withdrawal Period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ixekizumab | Placebo
Number analyzed (Participants) | 51 | 22
score on a scale | -0.79 (0.06) | -0.67 (0.06)

ADVERSE EVENTS:
Time Frame: Up To 3 Years
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- IXE80Q2W Non-randomized Population to Withdrawal Period: Participants completed open label but did not meet criteria for randomization to the double-blind Withdrawal Period.
  Participants continued to receive 80 mg given as one SC injection every two weeks during the double-blind withdrawal period.
- IXE80Q2W Relapse Period: IXE80Q2W Relapse Period
  Double Blind Period: 80 mg ixekizumab given as one SC injection Q2W from randomization to week 104 (or, early termination or relapse).
  Double Blind Period: Placebo given as one SC injection Q2W any time from randomization to week 104 (or, early termination or relapse).
Arm/Group | Ixekizumab Open Label | Ixekizumab | Placebo | IXE80Q2W Non-randomized Population to Withdrawal Period | IXE80Q2W Relapse Period | IXE80Q2W Post-Treatment Follow-up Period | Placebo Post-Treatment Follow-up Period
All-Cause Mortality (participants affected / at risk) | 2/394 | 0/79 | 0/79 | 0/133 | 0/97 | 0/355 | 0/12
Serious Adverse Events (participants affected / at risk) | 20/394 | 1/79 | 2/79 | 6/133 | 1/97 | 4/355 | 0/12
Other Adverse Events (participants affected / at risk) | 143/394 | 25/79 | 14/79 | 37/133 | 30/97 | 19/355 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab Open Label (N=394) | Ixekizumab (N=79) | Placebo (N=79) | IXE80Q2W Non-randomized Population to Withdrawal Period (N=133) | IXE80Q2W Relapse Period (N=97) | IXE80Q2W Post-Treatment Follow-up Period (N=355) | Placebo Post-Treatment Follow-up Period (N=12)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/212 (1) | 0/32 (0) | 0/39 (0) | 0/78 (0) | 0/53 (0) | 0/195 (0) | 0/6 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0/212 (0) | 1/32 (1) | 0/39 (0) | 0/78 (0) | 0/53 (0) | 0/195 (0) | 0/6 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/212 (0) | 0/32 (0) | 0/39 (0) | 1/78 (1) | 0/53 (0) | 0/195 (0) | 0/6 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab Open Label (N=394) | Ixekizumab (N=79) | Placebo (N=79) | IXE80Q2W Non-randomized Population to Withdrawal Period (N=133) | IXE80Q2W Relapse Period (N=97) | IXE80Q2W Post-Treatment Follow-up Period (N=355) | Placebo Post-Treatment Follow-up Period (N=12)
Injection site reaction (General disorders) | 59 (270) | 1 (8) | 0 (0) | 2 (20) | 7 (27) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 18 (23) | 4 (4) | 1 (1) | 5 (5) | 4 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 34 (37) | 11 (13) | 4 (4) | 19 (22) | 13 (17) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 9 (10) | 4 (9) | 1 (3) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 49 (66) | 9 (14) | 4 (5) | 12 (18) | 9 (10) | 8 (8) | 0 (0)
Alanine aminotransferase increased (Investigations) | 11 (14) | 4 (4) | 1 (2) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 4 (4) | 1 (2) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/212 (0) | 2/32 (2) | 0/39 (0) | 0/78 (0) | 0/53 (0) | 0/195 (0) | 0/6 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Statistical Analysis Plan: Statistical Analysis Plan V3 (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT02584855/SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Blinding and Unblinding Plan V3 (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02584855/SAP_001.pdf
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02584855/Prot_002.pdf